CLINICAL TRIAL: NCT04357184
Title: Blood Flow Restriction Training for Severe Lower Extremity Muscle Atrophy
Brief Title: BFRT for Severe Lower Extremity Muscle Atrophy
Acronym: BFRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cincinnati Sportsmedicine Research and Education Foundation (Other)
Responsible Party: Principal Investigator, Sue Barber-Westin, Director Clinical Studies, Cincinnati Sportsmedicine Research and Education Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFRT17-37
Record Dates: First submitted 2020-04-14; First posted 2020-04-22 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Severe Muscle Atrophy; Muscle Weakness
MeSH Terms: conditions — Muscular Atrophy; Muscle Weakness | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BFRT with 4 exercises and low resistance loads (Experimental): Blood flow resistance training will be performed with a standard blood pressure cuff that is placed and inflated by a clinician. The patient will perform 4 exercises with low resistance loads that will produce a muscle burn to enhance promotion of strength. Training will be supervised in the clinic. The cuff is deflated between exercises.
  Interventions: Other: Blood flow restriction training

INTERVENTIONS:
Other: Blood flow restriction training — BFRT is done with 4 exercises with low load resistance of 30% 1 repetition maximum

SUMMARY:
Muscle weakness or atrophy is a common condition following acute and chronic musculoskeletal injuries. Strength training is an imperative component in clinical rehabilitation of musculoskeletal injuries. Heavy exercise loads (approximately 70% of one repetition maximum) is necessary to elicit muscle hypertrophy and strength gains. However, patients with severe muscle atrophy are frequently unable to tolerate these loads due to pain. Blood flow resistance training with low resistance loads may be used to safely develop muscle strength.

DETAILED DESCRIPTION:
Blood flow restriction training (BFRT) is a safe type of low intensity resistance exercise that has demonstrated enhanced muscle growth, muscle strength, oxygen delivery and utilization (VO2Max). With BFRT, lighter loads can be used to build muscle while sparing the joints from heavy loading and without overly fatiguing the central nervous system.

The objectives of BFRT are 1) to increase the effectiveness of physical therapy, 2) safely increase muscle mass, reduce arterial stiffness, increase bone density, increase Vo2Max, improve carotid arterial compliance and enhance response of the autonomic nervous system, 3) improve muscle endurance in 1/3 the time, improve strength and hypertrophy after surgery, improve muscle recruitment and increase anabolic growth signaling.

ELIGIBILITY:
Inclusion Criteria:

* Patients with > 20% deficit in isometric quadriceps and/or hamstrings strength
* Patients willing to complete at least 9 BFRT training sessions
* Patients willing to provide informed consent (or parental consent)

Exclusion Criteria:

* Pregnancy
* History of varicose veins
* History of blood clots or active blood clot
* Taking oral contraceptives
* History of heart attack
* Unstable cardiac disease
* Taking heart failure medication
* Uncontrolled hypertension (> 140/90)
* Uncontrolled tachycardia (> 100 bpm)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Isometric quadriceps and hamstrings muscle strength | Strength will be measured for each patient before training begins and then after 9 training sessions have been completed, for the duration of the study, up to 100 weeks
  Isometric knee flexor and extensor strength will be measured with an isokinetic dynamometer before training and after each series of 9 training sessions

SECONDARY OUTCOMES:
Patient rating | The intensity of muscle burn will be determined during each training session. The overall satisfaction will be determined after the last training session for each patient, for the duration of the study, up to 100 weeks.
  Patients will rate the intensity of muscle burn produced during training and overall satisfaction with the final result

CONTACTS AND LOCATIONS:
Overall Officials: Frank R Noyes, MD, Principal Investigator — Cincinnati Sportsmedicine Research and Education Foundation
Locations (1):
- Cincinnati Sportsmedicine and Orthopaedic Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No